CLINICAL TRIAL: NCT01620099
Title: Small Airways Involvement in Smoker Asthmatic Patients: a Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, Alberto Papi, MD, Professor, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SAISA01
Record Dates: First submitted 2012-05-09; First posted 2012-06-15 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Asthma
Keywords: Asthma; Cigarette smoke; Small airways; Lung function; Asthma control
MeSH Terms: conditions — Asthma; Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asthmatic nonsmokers (Experimental): Asthmatic patients aged 18-50 years old, at stage 2-3 according to GINA international guidelines, on inhaled treatment (ICS alone or combination ICS/LABA) other than extrafine formulations, will be enrolled. This group includes patients who never smoked. Following the initial evaluation (cross-sectional - primary outcome) patients will be switched to an extrafine equipotent dose of the same compound (BDP-HFA if the patient was on ICS) or combination (BDP-HFA/F if the patient was on ICS/LABA combination). After 3-months patients will be reassessed for lung function and asthma control
  Interventions: Drug: Extrafine treatment (Clenilexx(R) or Foster(R))
- Asthmatic smokers (Active Comparator): Asthmatic patients aged 18-50 years old, at stage 2-3 according to GINA international guidelines, on inhaled treatment (ICS alone or combination ICS/LABA) other than extrafine formulations, will be enrolled. This group includes patients who smoked with a smoking habit ranging from 10 to 20 pack/years. Following the initial evaluation (cross-sectional - primary outcome) patients will be switched to an extrafine equipotent dose of the same compound (BDP-HFA if the patient was on ICS) or combination (BDP-HFA/F if the patient was on ICS/LABA combination). After 3-months patients will be reassessed for lung function and asthma control
  Interventions: Drug: Extrafine treatment (Clenilexx(R) or Foster(R))

INTERVENTIONS:
Drug: Extrafine treatment (Clenilexx(R) or Foster(R)) — Following the initial evaluation (cross-sectional) patients will be switched to an extrafine equipotent dose of the same compound (extrafine beclomethasone dipropionate - Clenilexx(R) - if the patient was on ICS) or combination (extrafine beclomethasone dipropionate/formoterol - Foster(R) - if the patient was on ICS/LABA combination). After 3-months patients will be reassessed for lung function and asthma control

SUMMARY:
Asthma is an inflammatory disease affecting the whole respiratory system, from central to peripheral airways. Anti-inflammatory treatment with inhaled corticosteroids (ICS), with or without long-acting β2-adrenoceptor agonists (LABA), is the cornerstone of asthma management [GINA Guideline - available at www.ginasthma.com]. Nevertheless, a considerable subset of asthmatic patients neither benefits from ICS nor gain optimal asthma control even with ICS/LABA combinations.

The involvement of the distal lung, i.e. the peripheral membranous bronchioles < 2 mm in diameter (so-called small airways), in the pathogenesis of asthma has been extensively investigated and its significance debated. However, whether specifically targeting distal lung abnormalities can lead to further clinical benefit is still an open question. In this context, interest has been raised by hydrofluoroalkane (HFA) pressurised metered-dose inhalers, which can deliver compounds with a mass median aerodynamic diameter that is significantly smaller than other available devices, leading to increase peripheral airways drug deposition.

Up to 30% of asthmatic patients smoke, mirroring the rate found in the general population. Several data document that smoking habit negatively affect corticosteroid efficacy in asthma. In particular, asthmatic patients who smoke experience faster lung function decline, increased frequency of exacerbations and reduced asthma control despite being regularly treated. Several molecular mechanisms have been proposed to address the issue of reduced corticosteroids responsiveness in smoker patients. However it has been never investigated whether reduced corticosteroid responsiveness in asthmatic patients who smoke can be related to more severe small airways involvement leading to impaired distribution or impaired peripheral deposition of inhaled corticosteroids. If this is the case, asthmatic patients who smoke might benefit from a pharmacological approach able to target and to reach small airways.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-50 years old, at stage 2-3 according to GINA international guidelines
* patients must be free from an exacerbation from at least 2 months
* patients must be on inhaled treatment (ICS alone or combination ICS/LABA) other than extrafine formulations from at least 3 months.
* according to smoking habit, patients will be divided in two groups:

  1. nonsmokers: patients who never smoked
  2. smokers: patients with a smoking habit ranging from 10 to 20 pack/years.

Exclusion Criteria:

* to avoid possible overlapping with chronic obstructive pulmonary disease, patients will not be included in the study if any of the following exclusion criteria are present:

  * aged > 50 years
  * heavy-smoker patients (pack/years > 20)
  * patients with a not fully reversible airflow obstruction (i.e. post-bronchodilator FEV1/FVC < 70%)
  * patients with an impaired diffusion capacity (DLCO < 80%v predicted).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
slope of phase III (dN2) by nitrogen single breath test | At baseline
  The primary outcome will measure and compare at baseline slope of phase III (dN2) by nitrogen single breath test (NSBT) between asthmatic who smoke and asthmatic who do not smoke matched for age, gender and % predicted FEV1

SECONDARY OUTCOMES:
Closing volume and closing capacity by nitrogen single breath test (NSBT) | At baseline
  To evaluate and compare at baseline other nitrogen single breath test measures including closing volume and closing capacity in asthmatic who smoke and asthmatic who do not smoke matched for age, gender and % predicted FEV1.
Respiratory Resistance by oscillometry technique | At baseline
  To evaluate differences in mean resistive component of respiratory impedence (Rrs) and resistance at different frequency (Rr0, Rr5, Rr20) by forced oscillometry technique (FOT) at baseline between asthmatics who smoke compared to asthmatics who do not smoke matched for age, gender and % predicted FEV1.
Lung volumes | At baseline
  To evaluate differences in forced vital capacity (FVC), slow vital capacity/forced vital capacity ratio (SVC/FVC), residual volume (RV) and total lung capacity (TLC) at baseline between asthmatics who smoke compared to asthmatics who do not smoke matched for age, gender and % predicted FEV1.
Asthma control | At baseline
  To evaluate differences in parameters related to asthma control (Asthma Control Test scores, use of rescue medications) at baseline between asthmatics who smoke compared to asthmatics who do not smoke matched for age, gender and % predicted FEV1.
Correlations between small airway functional parameters and asthma control scores | At baseline
  To evaluate at baseline correlations between parameters related to asthma control (questionnaire scores, symptoms and use of rescue medications) and functional measurements
Changes after extrafine intervention | Change at 3 months vs baseline
  To evaluate changes in functional parameters and parameters related to asthma control in asthmatic patients who smoke compared to asthmatic patients who do not smoke after a 3-months extrafine inhaled treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Papi, MD, Principal Investigator — Università degli Studi di Ferrara
Locations (2):
- Hospital Grosshansdorf, Großhansdorf, Germany
- Research Centre on Asthma and COPD, University of Ferrara, Ferrara, Italy

REFERENCES:
- [Background] Bateman ED, Boushey HA, Bousquet J, Busse WW, Clark TJ, Pauwels RA, Pedersen SE; GOAL Investigators Group. Can guideline-defined asthma control be achieved? The Gaining Optimal Asthma ControL study. Am J Respir Crit Care Med. 2004 Oct 15;170(8):836-44. doi: 10.1164/rccm.200401-033OC. Epub 2004 Jul 15. PMID 15256389
- [Background] Contoli M, Bousquet J, Fabbri LM, Magnussen H, Rabe KF, Siafakas NM, Hamid Q, Kraft M. The small airways and distal lung compartment in asthma and COPD: a time for reappraisal. Allergy. 2010 Feb;65(2):141-51. doi: 10.1111/j.1398-9995.2009.02242.x. Epub 2009 Nov 11. PMID 19909298
- [Background] Hampel F, Lisberg E, Guerin JC. Effectiveness of low doses (50 and 100 microg b.i.d) of beclomethasone dipropionate delivered as a CFC-free extrafine aerosol in adults with mild to moderate asthma. Study Group. J Asthma. 2000 Aug;37(5):389-98. doi: 10.3109/02770900009055464. PMID 10983616
- [Background] Haussermann S, Acerbi D, Brand P, Herpich C, Poli G, Sommerer K, Meyer T. Lung deposition of formoterol HFA (Atimos/Forair) in healthy volunteers, asthmatic and COPD patients. J Aerosol Med. 2007 Fall;20(3):331-41. doi: 10.1089/jam.2007.0613. PMID 17894539
- [Background] Leach CL, Davidson PJ, Hasselquist BE, Boudreau RJ. Lung deposition of hydrofluoroalkane-134a beclomethasone is greater than that of chlorofluorocarbon fluticasone and chlorofluorocarbon beclomethasone : a cross-over study in healthy volunteers. Chest. 2002 Aug;122(2):510-6. doi: 10.1378/chest.122.2.510. PMID 12171824
- [Background] Thomson NC, Chaudhuri R. Asthma in smokers: challenges and opportunities. Curr Opin Pulm Med. 2009 Jan;15(1):39-45. doi: 10.1097/MCP.0b013e32831da894. PMID 19077704
- [Background] Chalmers GW, Macleod KJ, Little SA, Thomson LJ, McSharry CP, Thomson NC. Influence of cigarette smoking on inhaled corticosteroid treatment in mild asthma. Thorax. 2002 Mar;57(3):226-30. doi: 10.1136/thorax.57.3.226. PMID 11867826
- [Background] Tomlinson JE, McMahon AD, Chaudhuri R, Thompson JM, Wood SF, Thomson NC. Efficacy of low and high dose inhaled corticosteroid in smokers versus non-smokers with mild asthma. Thorax. 2005 Apr;60(4):282-7. doi: 10.1136/thx.2004.033688. PMID 15790982
- [Background] Pedersen SE, Bateman ED, Bousquet J, Busse WW, Yoxall S, Clark TJ; Gaining Optimal Asthma controL Steering Committee and Investigators. Determinants of response to fluticasone propionate and salmeterol/fluticasone propionate combination in the Gaining Optimal Asthma controL study. J Allergy Clin Immunol. 2007 Nov;120(5):1036-42. doi: 10.1016/j.jaci.2007.07.016. Epub 2007 Nov 1. PMID 17935765
- [Background] Chapman KR, Boulet LP, Rea RM, Franssen E. Suboptimal asthma control: prevalence, detection and consequences in general practice. Eur Respir J. 2008 Feb;31(2):320-5. doi: 10.1183/09031936.00039707. Epub 2007 Oct 24. PMID 17959642
- [Background] Adcock IM, Caramori G, Ito K. New insights into the molecular mechanisms of corticosteroids actions. Curr Drug Targets. 2006 Jun;7(6):649-60. doi: 10.2174/138945006777435344. PMID 16787166
- [Derived] Contoli M, Bellini F, Morandi L, Forini G, Bianchi S, Gnesini G, Marku B, Rabe KF, Papi A. Assessing small airway impairment in mild-to-moderate smoking asthmatic patients. Eur Respir J. 2016 Apr;47(4):1264-7. doi: 10.1183/13993003.01708-2015. Epub 2016 Feb 11. No abstract available. PMID 26869674